CLINICAL TRIAL: NCT07165366
Title: Clinical Evaluation of Enamel Microhardness Using At-Home and In-Office Tooth Whitening Agents
Brief Title: Clinical Evaluation of Enamel Microhardness Using Tooth Whitening Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ultradent Products, Inc. (Industry)
Collaborators: Universidad Intercontinental (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1-2025 Enamel Hardness
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Dental Atraumatic Restorative Treatment
Keywords: enamel loss; demineralization

STUDY DESIGN:
Intervention Model Description: In the mouth there are two bicuspids in each quadrant. One bicuspid in the maxillary arch was treated with 10% CP for 14 days. One bicuspid in the mandibular arch was treated with 40% HP. The other bicuspids in the other two quadrants were untreated, negative controls.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Teeth left untreated as control group.
- OP 10% CP (Experimental): Teeth treated with 10% CP over a14 day span
  Interventions: Diagnostic Test: Carbamide Peroxide 10%
- OP 40% HP (Experimental): Teeth treated with 40% Hydrogen Peroxide
  Interventions: Diagnostic Test: Hydrogen Peroxide

INTERVENTIONS:
Diagnostic Test: Carbamide Peroxide 10% — treatment over 14 days of 10% Carbamide Peroxide
  Arms: OP 10% CP
Diagnostic Test: Hydrogen Peroxide — treatment of 40% Hydrogen Peroxide
  Arms: OP 40% HP

SUMMARY:
The investigator will review the medical history taken by the participants' orthodontist that determined participants eligibility to participate in this study on the first appointment. If the investigator determines that the position and condition of participants' teeth meet the inclusion and exclusion criteria for participation in this study, the participant will be enrolled to participate in the study. Once accepted, a small area (1 mm) of the premolars will be flattened and polished. Next, participants upper teeth will be scanned to make an impression, and the bleaching tray will be made on it. None of these procedures are painful, nor do they require anesthesia. This first appointment will last about 60 minutes. At the second appointment, the initial color of the upper premolar to be bleached will be taken. Participants will also be given a personalized whitening tray, a container to store the tray when not in use, a tube of low-concentration teeth whitening agent, and a toothbrush and toothpaste. The investigator will show participants how to place the tray on the upper arch. Participants will wear it through the night for fourteen nights. Participants will be given a chart to mark every night when the tray is used and teeth are brushed. Investigators will call participants the next day and in 7 days to see if participants have had any problems putting the gel in the tray and using it. This appointment will last approximately 30 minutes. The third appointment will consist of the investigator isolating one of the lower premolars that will be extracted. Some gel will be applied to that tooth three times; each time, the gel will stay on participant's tooth for 20 minutes. If the soft tissue or tooth is sensitive, a soothing gel will be applied to relieve the discomfort. This appointment will last approximately 90 minutes. The fourth appointment will be 14 days after the at-home bleaching was done and the in-office bleaching was accomplished. During this appointment, a lower premolar might be etched for 15 seconds. At this appointment, the oral surgeon the participant's orthodontist recommends will extract the participant's teeth. That will be the final appointment. During these 14 days, participant must keep cleaning teeth every day at least twice a day.

DETAILED DESCRIPTION:
14- PROJECT METHODOLOGY: Methods and materials This study consists of 40 patients requiring the extraction of four permanent first or second premolars for orthodontic reasons. Patients will be recruited from the Universidad Intercontinental (UIC) Graduate Program in Orthodontics, and private orthodontist dental offices in the city of Mexico. Patients who identify as needing extraction of the four first or second permanent premolars and who meet the following inclusion criteria will be invited to participate in the study.

Inclusion criteria:

* Have the four premolars in different quadrants that their orthodontist recommends be extracted.
* The premolars to be extracted should have prominent facial surfaces.
* Willing to have the four premolars slightly flattened and smoothed.
* Willing to have all four premolars extracted for orthodontic reasons.
* Between 12 and 35 years of age.
* Willing to attend four appointments.
* Willing to wear a custom-made whitening tray during the evening when they sleep.
* Willing to have their premolars bleached with In-Office and At-Home bleaching agents and one of their teeth that will be extracted treated with phosphoric acid.
* Willing to sign a consent form (parents must co-sign if they are under 18).
* Willing to discontinue active orthodontic treatment during whitening treatment.
* Willing to brush at least twice a day with fluoridated toothpaste provided during the study.

Exclusion criteria:

* Restorations or visible cavities in any tooth to be extracted.
* The presence of visible intraoral structural defects or pathology.
* Use of over-the-counter or professionally prescribed whitening agents in the past six months.
* Teeth with tetracycline staining.
* History of any medical illness that may interfere with the study or require special considerations.
* Pregnant or lactating women.
* Not willing to do the blood tests (biometrics hematic, prothrombin, and thromboplastin) prior to extractions (a legal requirement of the Oral Surgery Department of the UIC).

Treatment plan:

The study will be approved by Ultradent Products, Inc. and the Health Sciences Divisional Area Bioethics Committee, which is the equivalent of the Institutional Review Board (IRB) of UIC before any patients will be evaluated for eligibility to enter the study.

At the first appointment (selection appointment), the absence of evident cavities or restorations in the four premolars will be clinically verified with an intraoral mirror. Root formation will be confirmed with the panoramic radiograph from the patient's orthodontic chart. The treatment will be explained, and the patient will be allowed to ask questions and discuss any concerns. Subjects will be informed that the study will consist of 4 appointments. If the patient qualifies and agrees to be part of the study, they will be asked to sign an approved Consent Form. Parents or guardians will be asked to sign the consent form for patients under 18 years of age. Participants will be given a copy of the signed Consent Form. The requirements are that the four teeth that will be extracted for orthodontic reasons will be flattened and polished to produce a one-by-one millimeter surface on the facial or most prominent surface. This will be done with a 169L bur and fine and extra-fine sandpaper discs. Additionally, they must agree to use a whitening tray every night for 14 nights with Opalescence 10% CP with or without PF (potassium nitrate and fluoride) on an upper right premolar (UR) or on the upper left premolar (UL) (the tooth that has the best alignment). The contralateral lower right (LR) or lower left (LL) premolar will be treated with 40% hydrogen peroxide (HP) Opalescent Boost PF at the dental clinic for three 20-minute periods according to the manufacturer's instructions**. Thirty of the 40 subjects will treat their UR or UL premolar treated with Opalescence 10% CP with PF. The remaining 10 subjects will treat their UR or UL premolar with Opalescence 10% CP without PF.

A digital scan impression (Dentsply Sirona Scanner) of each subject's dentition will be taken and study models fabricated. On the UR or UL premolar of the model, a 0.5 mm thick resin veneer of unfilled Block-Out-Resin (Ultradent Products Inc.) will be placed. The veneer will be applied on the facial surface or, by exception, on the lingual surface (the most prominent) of the tooth at 1.0 mm mesial, distal, and incisal, and 1.5 mm from the gingival margin. The resin veneer will be light-cured for 15 seconds using a standard visible curing light unit. Bleaching trays will be fabricated from 0.035-inch plastic sheets (Sof-Tray; Ultradent Products Inc.) on each subject's digital model and appropriately trimmed in the UIC laboratory and/or in a private practice laboratory. The trays will be trimmed with microscissors, 0.5 mm from the gingival margin. If the patient has started the placement of braces and/or orthodontic bands, the trays will be modified with "windows" to accommodate the brackets, if necessary, and the second molars in the bleaching trays will be removed to allow a better adaptation (no movements or orthodontic treatments will be allowed in any of the four premolars to be extracted).

The second appointment will occur at least 24 hours after the first appointment. The subject will receive the maxillary whitening tray with a single reservoir for the UR or UL premolar, a tube of Opalescent 10% CP containing or not containing PF whitening gel, and a container for tray storage, when tray is not in use. During this appointment, the color of that premolar will be taken with VITA Bleachedguide 3-D MASTER shade guide (VITA, Zahnfabrik, Germany). The tray will be placed in the mouth to ensure a proper fit without interference. The subject will be instructed to place a small amount of whitening gel into the individual reservoir for the UR or UL premolar each evening, then carefully placing the tray over the teeth, and wipe off the excess gel. The subject will be instructed to wear the bleaching tray for at least 8 hours every night, for 14 nights, after brushing their teeth. Each morning after using the tray, the subject will be instructed to brush off the used gel, rinse the tray, store it in the container provided, and brush their teeth with the toothpaste provided. Subjects need to brush thoroughly twice a day, morning and night. During the 14 days of whitening at home, the subject will be contacted twice by phone or text message to make sure they are using the tray with the whitening gel, properly.

The third appointment will occur on day 15. The subject will return the maxillary whitening tray and will be encouraged to report any concerns with the bleaching treatment or tray usage. During this appointment, the LR or LL premolar and collateral to the premolar that was bleached at-home will be isolated with OpalDam (Ultradent Products, Inc.) and will be treated with Opalescent Boost 40% HP. The treatment will consist of application of the gel three separate times, each for will remain on the one premolar for 20 minutes, according to the manufacturer's instructions*. If the soft tissue or tooth becomes sensitive, a soothing gel will be applied to relieve discomfort (Opalescence UltraEZ). Tissue sensitivity usually lasts about thirty minutes and tooth sensitivity usually decreases in two or three days. This appointment will last approximately 90 minutes. During this appointment, an orthodontic separator band or elastic band of 2.5 to 4.5 oz / ⅛" to ¼" (depending on interproximal access) will be placed in the gingival area of each premolar to create bone resorption and facilitate an atraumatic extraction. The final color will be taken of the premolar that received 14 days of whitening at-home, as well as the initial and final color of the premolar that will be bleached in-office with VITA Bleachedguide 3-D Master (VITA Zahnfabrik); this is to corroborate and document that the teeth were successfully whitened. At this appointment, the subject will be reminded to complete the blood tests required by the UIC oral surgery department since, without these lab tests, the extractions cannot be performed. Therefore, the compensation would not be completed. Also, the subject will be reminded to continue documenting on the log the brushing of at least twice a day for at least one minute each time and will be asked to follow these instructions for the next 14 days.

The fourth and final appointment will take place on day 29, in other words,14 days after the third appointment and 14 days after they have already finished their whitening treatment at home and in the office. At this appointment, 6 subjects, three of the 30 subjects that used 10% CP with PF and three of the 10 subjects that used 10% CP without the PF, will have their mandibular second control tooth etched with 35% phosphoric acid (Ultradent Products, Inc.) for 15 seconds. These 6 subjects will be chosen to be treated before extractions with the etchant at a time convenient to the oral surgeon and Dr. Fugaro. Extractions will be performed during this appointment for all subjects. Four to five UIC maxillofacial surgeons will perform the extractions. Local anesthetics will be at the discretion of the oral surgeon and the patient's needs. Extractions will be performed with a simple elevator forceps technique as described in the attached protocol**. Immediately after extractions, the teeth will be cleaned to remove any debris with a dental curette without touching the treated area. The teeth will then be placed in a plastic snap top container (Fisher Scientific) with a wet sponge (sodium-free drinking water) and 0.12% chlorhexidine at the bottom of the bottle and snapped closed. Each vial will be labeled with the date of extraction, a subject identification number, the subject's initials, the tooth number, and how the tooth was treated (at home, in office, etched, or control) and forwarded for testing to Therametric Technologies, Inc.

ELIGIBILITY:
Inclusion criteria:

* Have the four premolars in different quadrants that their orthodontist recommends be extracted.
* The premolars to be extracted should have prominent facial surfaces.
* Willing to have the four premolars slightly flattened and smoothed.
* Willing to have all four premolars extracted for orthodontic reasons.
* Between 12 and 35 years of age.
* Willing to attend four appointments.
* Willing to wear a custom-made whitening tray during the evening when they sleep.
* Willing to have their premolars bleached with In-Office and At-Home bleaching agents and one of their teeth that will be extracted treated with phosphoric acid.
* Willing to sign a consent form (parents must co-sign if they are under 18).
* Willing to discontinue active orthodontic treatment during whitening treatment.
* Willing to brush at least twice a day with fluoridated toothpaste provided during the study.

Exclusion criteria:

* Restorations or visible cavities in any tooth to be extracted.
* The presence of visible intraoral structural defects or pathology.
* Use of over-the-counter or professionally prescribed whitening agents in the past six months.
* Teeth with tetracycline staining.
* History of any medical illness that may interfere with the study or require special considerations.
* Pregnant or lactating women.
* Not willing to do the blood tests (biometrics hematic, prothrombin, and thromboplastin) prior to extractions (a legal requirement of the Oral Surgery Department of the UIC).

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Matis, DDS, MSD, Principal Investigator — Indiana University
Locations (1):
- Universidad Intercontinental, Mexico City, Tialpan, Mexico

IPD SHARING:
Plan to Share IPD: No
We will share information after it is published.

REFERENCES:
- See also: Study Protocol — https://indiana-my.sharepoint.com/:w:/g/personal/tmatis_iu_edu/EXk1Wua2GxBPo1gcO7KMZxUBEu5I3HUln-A2paATQIxsOg?e=Zdtd69
- Available data/document: Informed Consent Form — https://indiana-my.sharepoint.com/:w:/g/personal/tmatis_iu_edu/EalUzspTf7VClbHYAyBlJg4BVp2wl1gK8uHn7MzUbZ4tbA?e=1vfYnE
- Available data/document: Statistical Analysis Plan — https://indiana-my.sharepoint.com/:w:/g/personal/tmatis_iu_edu/EbDir0nT8JNAlpv4-vfnOxMBCBxsvrV2UjY2_ua4APTs2g?e=zJdPmF

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients at the Postgraduate Department of Orthodontics at the Universidad Intercontinental were invited to participate in the study. The recruitment period began on May 1,2024
Pre-assignment Details: Participants were excluded who did not have prominent facial surfaces on a bicuspid in each of their four quadrants.
Units Other Than Participants: teeth
Groups:
- Control: Teeth in patients that were left untreated during the trial. (2 units)
- OP 10% CP: Teeth in patients that were exposed to 10% Carbamide Peroxide over a consecutive 14-day period. (1 unit)
- OP 40% HP: Teeth in patients that were exposed to 40% Hydrogen Peroxide in a single session.(1 unit)
Period: Overall Study
Arm/Group | Control | OP 10% CP | OP 40% HP
Started | 40; 80 teeth | 40; 40 teeth | 40; 40 teeth
Completed (Forty participants were utilized for this study, and each participant had four pre-molars set as either of untreated (two as control), treated with 10% CP or treated with 40% HP.) | 40; 80 teeth | 40; 40 teeth | 40; 40 teeth
Not Completed | 0; 0 teeth | 0; 0 teeth | 0; 0 teeth

BASELINE CHARACTERISTICS:
Population: Forty participants in total were utilized for the study. Each participant had 4 pre-molars included as part of the study, broken down into 2 control, one OP 10% CP and one OP 40% HP . The microhardness change at baseline could not be measured. Only Vickers microhardness after extraction will be determined.
Units Other Than Participants: teeth
Groups:
- Control: Untreated teeth
- OP 10% CP: Teeth treated with 10% Carbamide Peroxide for 14 days
- OP 40% HP: Teeth treated once with 40% Hydrogen Peroxide
- Total: Total of all reporting groups
Arm/Group | Control | OP 10% CP | OP 40% HP | Total
Number analyzed (Participants) | 40 | 40 | 40 | 160
Number analyzed (teeth) | 80 | 40 | 40 | 160
Age, Continuous [Geometric Mean (Full Range); unit: years] — Population: The total of patients was 40. Being 4 premolars analyzed for each patient. 2 teeth served as control group without treatment, 1 for OP 10% CP; and 1 OP 40% HP.
  years
    number analyzed (Participants) | 40 | 40 | 40 | 40
    (all) | 18.7 [12 to 35] | 18.7 [12 to 35] | 18.7 [12 to 35] | 18.7 [12 to 35]
Sex: Female, Male [Count of Units; unit: teeth] — The total of patients was 40. Being 4 premolars analyzed for each patient. 2 teeth served as control group without treatment, 1 for OP 10% CP; and 1 OP 40% HP. Population: The total of patients was 40. Being 4 premolars analyzed for each patient. 2 teeth served as control group without treatment, 1 for OP 10% CP; and 1 OP 40% HP. The unit of measure was Vickers hardness of each teeth, measured on the buccal surfaces.
  teeth
    number analyzed (Participants) | 40 | 40 | 40 | 40
    Female | 52 | 26 | 26 | 104
    Male | 28 | 14 | 14 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0
    (all) |  |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Enamel Hardness
Description: Vickers hardness kg f/mm2
  Baseline measurements: two nonbleached bicuspids in the dental arches. One first or second bicuspid in the maxillary arch was bleached with At-Home 10% Carbamide Peroxide and the contralateral bicuspid served as the control in the maxillary arch. One first or second bicuspid in the mandibular arch was bleached with In-Office 40% Hydrogen Peroxide and the other contralateral bicuspid in the mandibular arch served as the control. The control bicuspids served as the baseline measurements.
Time Frame: one month
Population: Two teeth serve as control.
Measure: Mean (95% Confidence Interval); unit: Vickers hardness kg f/mm2
Units Other Than Participants: teeth
Groups:
- OP 10% CP: Teeth treated with 10% Carbamide Peroxide over a consecutive 14-day period.
- OP 40% HP: Teeth treated with 40% Hydrogen Peroxide in a single session.
Arm/Group | Control | OP 10% CP | OP 40% HP
Number analyzed (Participants) | 40 | 40 | 40
Number analyzed (teeth) | 80 | 40 | 40
Vickers hardness kg f/mm2 | 348.4 [342.0 to 354.7] | 351.6 [341.9 to 361.2] | 354.5 [346.8 to 362.3]
Statistical Analysis 1: Comparison: Control vs OP 10% CP vs OP 40% HP; Null Hypothesis is that there will be no difference in enamel hardness when different concentrations are used on enamel surfaces; Test type: Superiority; p = 0.231, ANOVA — a priori threshold for significance was alpha=0.05; degrees of freedom for ANOVA F-statistic were 2 for numerator d.f. and 118 denominator d.f; F-statistic = 1.48

ADVERSE EVENTS:
Time Frame: Patients were contacted twice during the 14 days of initial treatment time (Day 1 and day 7) . Patients did not report any unexpected discomfort. Patients were followed up for 30 days post treatment. There were no fatalities during the study.
Description: No serious adverse events were reported. Minor discomfort during extraction that occurred was expected.
Arm/Group | Control | OP 10% CP | OP 40% HP
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT07165366/Prot_000.pdf
  • Statistical Analysis Plan: statistical analysis plan (2024-04-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT07165366/SAP_001.pdf
  • Statistical Analysis Plan: Updated statistical analysis plan (2024-04-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT07165366/SAP_002.pdf
  • Informed Consent Form (2024-04-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT07165366/ICF_003.pdf